CLINICAL TRIAL: NCT01025414
Title: The Use of Enteral Nutrition in the Treatment of Pancreatic Fistulas - A Prospective, Randomized Clinical Trial
Brief Title: Enteral Nutrition in the Treatment of Pancreatic Fistulas - A Prospective Study
Acronym: FIS-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Stanislaw Klek MD PhD, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fistula-1; CMUJ-FIS-1 (Other: Jagiellonian University)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Pancreatic Fistula
Keywords: pancreatic fistula
MeSH Terms: conditions — Pancreatic Fistula | interventions — Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: enteral nutrition — Group A - enteral feeding was started 2 to 4 hours after catheter placement via enteral tube inserted via endoscope below the Treitz's ligament into first intestinal loop (location of the tip) (Nutricial Ltd. Flocare). The initial flow rate was 10 ml/ hour, final 125 ml/ hour. Energy requirements was calculated using following rule: 0.15-0.2 gN/ kg and 130-170 kcal/ gN. Diet: Peptisorb (Nutricia Ltd.) - oligopeptide diet well tolerated by intestines
  Other Names: Peptisorb, Nutricia Ltd, Netherlands
Drug: Parenteral nutrition — Parenteral nutrition was started 2 to 4 hours after venous catheter placement (standard Arrow type, the tip located 5 cm over right vestibule, the location confirmed on chest X-ray) and continued until oral diet covering at least 60% of daily caloric and protein demand. The energy requirements were calculated using following rule: 0.15-0.2 gN/ kg and 130-170 kcal/ gN. Parenteral diets: Aminoplasmal 10%, Lipofundin LCT/MCT 10 and 20%, 40% Glucose, Tracutil (microelements and trace elements), Cernevit (vitamins), electrolytes
  Other Names: intravenous feeding

SUMMARY:
The primary objective of this study is to evaluate the effectives of enteral nutrition in the treatment of pancreatic fistulas. The ratio of pancreatic fistula closure after 30 days is selected as the primary outcome measure with the null hypothesis assuming that enteral nutrition provides better results than parenteral nutrition as far as the closure ratio, time to closure and treatment-related complications are concerned.

DETAILED DESCRIPTION:
The research into field of the role of enteral nutrition in the treatment of pancreatic fistulas is fully justified by the lower cost and complications' rate of EN compared to PN observed in clinical trials comparing enteral and parnetral route of feeding in pre- and postoperative period. Such authors as Braga, Torosian, Lewis or Sand et al. proved that use of enteral nutrition led to smaller amount of complication (especially infectious) and improved the outcome of surgery. The only method to verify the role of enteral nutrition is the prospective, randomized clinical trial.

STUDY OBJECTIVES 2.1 Primary Objective The primary objective of this study is to evaluate the effectives of enteral nutrition in the treatment of pancreatic fistulas. The ratio of pancreatic fistula closure after 30 days is selected as the primary outcome measure with the null hypothesis assuming that enteral nutrition provides better results than parenteral nutrition as far as the closure ratio, time to closure and treatment-related complications are concerned.

2.2 Secondary Objectives

The secondary objectives are to:

* determine time to fistula closure (defined as time between initiation of treatment and confirmed fistula closure),
* determine rates of fistula and treatment-related complications,
* assess changes in quality of life (QoL),
* determine economic costs of therapy. (for such terms as: fistula closure, time to closure see definition on page 3) For QoL assessment the EORTC QLQ - PAN26 score in Polish version (translation was approved by EORTC) will be used.

Benefits of the study:

1. the implementation of safer and less expensive conservative procedure. Basis: Costs of enteral nutrition are significantly lower than PN and EN is significantly safer than PN especially as far as infectious complications are concerned.
2. the enhancement of indications for enteral nutrition.

The confirmation of the null hypothesis allows recommending enteral nutrition as a method of choice for pancreatic fistula treatment.

ELIGIBILITY:
Inclusion Criteria:

* the presence of pancreatic fistula (PF) (verification of serum lipase concentration in drained fluid, findings on imaging modalities: endoscopic retrograde cholangiopancreatography (ERCP), helical computed tomography(hCT), magnetic reissonance imaging (MRI), ultrasonography (USG) or intraoperative surgeon's verification - any or some or all of them)
* good general status (Karnoffsky > 80, Eastern Cooperative Oncology Group (ECOG) scale 0 or 1; see Appendix 2);
* NRS and MUST evaluation - low/ medium risk patients not requiring parenteral nutrition as the essence treatment option,
* no PF's complication requiring special treatment present, such as intraabdominal abscess formation, pleuropneumonia, bleeding, paralytic ileus, etc. Complications will be diagnosed and treated according to generally accepted medical knowledge, standards and procedures.
* age below 80 and over 18;
* in case of neoplastic patients: no confirmed neoplastic dissemination nor distant metastases;
* no severe concomitant disease (heart failure, COPD, CABG, etc.);
* no history of known allergies or drug intolerance;
* informed consent

Exclusion Criteria:

* PF diagnosis uncertain;
* poor general status (Karnoffsky <80, ECOG > 1);
* the presence of serious complications; see above
* recent history of severe heart, lung, kidney or liver failure;
* the history of allergies or drug intolerance;
* confirmed neoplastic spread;
* severe malnutrition requiring combined treatment (PN+EN)
* withdrawal of consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The ratio of pancreatic fistula closure after 30 days is selected as the primary outcome measure | 30 days

SECONDARY OUTCOMES:
Rates of fistula and treatment-related complications, changes in quality of life | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, MD PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Nutrimed Medical Corporation, Krakow, Malopolska, Poland

REFERENCES:
- [Derived] Klek S, Sierzega M, Turczynowski L, Szybinski P, Szczepanek K, Kulig J. Enteral and parenteral nutrition in the conservative treatment of pancreatic fistula: a randomized clinical trial. Gastroenterology. 2011 Jul;141(1):157-63, 163.e1. doi: 10.1053/j.gastro.2011.03.040. Epub 2011 Mar 24. PMID 21439962